CLINICAL TRIAL: NCT05177146
Title: Neural Correlates of Anti-suiciDal rEsponse to kEtamine in Treatment Resistant biPolar dePression (DEEPP-Study)
Brief Title: Neural Correlates of Ketamine's Anti-suicidal Effects in Bipolar Depression
Acronym: DEEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 179-2020
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Bipolar Disorder (BD); Suicidality
Keywords: Transcranial magnetic stimulation (TMS); Open-label trial; Pilot study; Ketamine; Intravenous drug delivery (IV); N-methyl-d-aspartate (NMDA); Receptor antagonist; Electromyography (EMG); Electroencephalography (EEG); Intra-cortical facilitation (ICF); Short-interval cortical inhibition (SICI)
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Ketamine (IV) (Experimental)
  Interventions: Drug: Intravenous Ketamine (IV)

INTERVENTIONS:
Drug: Intravenous Ketamine (IV) — A sterile form of ketamine hydrochloride will be administered over 40-min IV infusion twice per week on non-consecutive days for four weeks. Dosing schedule is determined based on patient's weight, clinical response and tolerability. First treatment session dose will be calculated based on 0.5 mg/kg. Further dose increase will be determined by the study physician. Dose increase will not exceed 0.8 mg/kg. Patients will be closely monitored by available trained personnel with MD being present on site for the full duration of the 2-h supervision period. Specifically, IV induction will be performed under the direct supervision of anesthesiologist or delegate and psychiatrist. Vital signs will be monitored every 30 minutes during the supervision period. Side effects will be managed by the medical team administering the treatment. If required, appropriate rescue medications will be provided depending on the nature of the adverse event.

SUMMARY:
Bipolar disorder is characterized by manic episodes and episodes of extreme depressive feelings, also known as bipolar depression (BD). Although clinical data does not suggest significant differences in the severity of depressive symptoms between bipolar and unipolar depression, patients with BD are found to be more likely to experience suicidal ideation and suicide attempts. Innovative treatments for suicidality in patients with BD are needed to address tolerability and slow effect limitations of current interventions. Using an open label pilot study, this trial aims to examine the effect of Intravenous (IV) ketamine treatment on acute suicidality in patients with BD. Moreover, the study aims to explore the neurophysiological mechanisms of ketamine's action directly from the cortex in patients with BD, in order to understand the biological mechanism underlying ketamine's therapeutic action.

DETAILED DESCRIPTION:
Ketamine is a fast-acting anesthetic that can have stimulant effects when taken at low doses. It acts as a non-competitive high-affinity N-methyl-d-aspartate (NMDA) receptor antagonist that stimulates synaptic glutamate release and blocks extra-synaptic NMDA receptors. This mechanism of action mediates excitatory synaptic transmission through the central nervous system and therefore results in robust antidepressant effects. Sub-anesthetic doses of ketamine administered intravenously (IV) have shown to produce rapid antidepressant and ant-suicidal effects. Despite this important clinical finding, our understanding of ketamine's neurophysiological mechanism of action for suicidality remains limited. This clinical trial is an open label pilot study that aims to address this limitation by studying the effects of IV ketamine on patients with bipolar depression who are currently experiencing suicidal thoughts. Using a combination of Transcranial Magnetic Stimulation (TMS) neurophysiological tools with electromyography (EMG) and electroencephalography (EEG), this trial aims to explore ketamine's action on NMDA neurotransmission to understand ketamine's anti-suicidal effects. Investigating the impact of ketamine on cortical excitation, cortical inhibition, and resting-state cortical oscillation could provide insight into the role of NMDA receptors in cortical physiology and determine potential predictors of clinical response for suicidality in bipolar depression.

Objective 1: To examine the effect of a series of therapeutic IV ketamine 40-min infusions on neurophysiological markers linked with cortical excitation and inhibition (as indexed via TMS-EMG and TMS-EEG, as a proxy of NMDA-receptor activity in the cortex)

Hypothesis 1: Ketamine will increase intracortical facilitation - a neurophysiological measure of NMDA neurotransmission

Objective 2: To examine the effect of ketamine IV 40-min infusions in sub-anesthetic doses on acute suicidality in patients with BD

Hypothesis 2: Ketamine infusions will result in improvement of suicidality in BD

Objective 3: To examine the safety and tolerability of ketamine IV 40-min infusions in sub-anesthetic doses and its effect on depressive symptoms in patients with BD

Hypothesis 3:

1. Ketamine infusions will be safe and well tolerated
2. Ketamine infusions will result in improvement of depressive mood symptoms in BD

Objective 4: To examine the effect of ketamine IV 40-min infusions in sub-anesthetic on additional neurophysiological measures and on changes in quality of life measures

Hypothesis 4:

1. Ketamine will decrease cortical inhibitory measures as indexed by (SICI) paradigms
2. Ketamine will increase cortical excitation measures as indexed by TMS-evoked potential waveform amplitude
3. Ketamine infusions will result in improvement in quality of life measures

ELIGIBILITY:
Inclusion Criteria:

1. Individual meeting DSM-IV diagnostic criteria for Bipolar Disorder, current depressive episode as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
2. Individuals capable to provide consent and able to communicate, read and write in English
3. Individuals currently depressed defined as scoring 14 and above on the Hamilton Rating Scale for Depression-24 Items (HRSD-24)
4. Individuals currently experiencing suicidal ideation as defined by a score of 9 or higher on the scale for suicide ideation (SSI)

Exclusion Criteria:

1. Individuals with history of a DSM-IV substance use disorder (i.e. dependence or abuse) within the past month; and lifetime history of ketamine substance use disorder as confirmed by the MINI
2. Concomitant major unstable medical illness such as poorly controlled high blood pressure or patients diagnosed with enlarged prostate or reporting any other urinary related issues
3. Stage 2 hypertension defined as a systolic pressure of 140 mm Hg or higher or a diastolic pressure of 90 mm Hg or higher on three consecutive readings taken 5 minutes apart
4. Results of liver function tests (ALT, AST) are three times or greater than the upper limit of normal readings
5. Pregnancy or the intention to become pregnant and breastfeeding during the study as confirmed by self-report. Female participants of reproductive potential must be willing to use a medically acceptable method of birth control which include highly effective (e.g. approved hormonal contraceptives, IUD, tubal ligation) or double barrier (e.g. male condom with diaphragm, male condom with cervical cap) methods of contraception or abstinence if that is the usual and preferred lifestyle of the participant
6. Presence of cardiac decompensation/heart failure
7. DSM-IV diagnosis of any primary psychotic disorder, bipolar disorder, obsessive-compulsive disorder, or post-traumatic stress disorder (current) as confirmed by the MINI
8. Current episode meeting criteria for mania/hypomania or mixed episode as per DSM-IV criteria on the MINI or as determined by the study team
9. Diagnosis of severe personality disorder as assessed during the initial consultation with a physician at the Temerty Centre prior to study entry
10. Any significant neurological disorder (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis) as assessed through medical history review during the initial consultation with a physician at the Temerty Centre prior to study entry
11. Individuals presenting with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator
12. Individuals requiring a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher; being on any anticonvulsant(e.g. Lamotrigine) and/or opioid medication due to the potential of these medications to limit the efficacy of ketamine
13. Individuals unable to communicate in spoken and written English fluently enough to complete the required study assessments due to a language barrier or a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete clinical assessments)
14. Individuals with cognitive or physical impairment which may potentially interfere with IN ketamine administration and subject's ability to stay in the same place for a 2-hr monitoring supervision as assessed through medical history review during the initial consultation with a physician at the Temerty Centre prior to study entry
15. Any intracranial implant (e.g., aneurysm clips, shunts, cochlear implants) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed given that we will be using TMS-EMG/EEG
16. Those unable to secure escort to accompany them back home after ketamine sessions will also be excluded from this study
17. Any known allergy to the study medication or any component/ingredient of the ketamine preparation

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Impact of a series of therapeutic IV Ketamine 40-min infusions on cortical excitation as measured by intracortical facilitation (ICF) | 1 month
  Assessed through administration of neurophysiological paradigms using Transcranial Magnetic Stimulation (TMS) paired with electromyography (EMG) and electroencephalography (EEG).
Impact of a series of therapeutic IV Ketamine 40-min infusions on cortical inhibition as measured by short-interval cortical inhibition (SICI) | 1 month
  Assessed through administration of neurophysiological paradigms using Transcranial Magnetic Stimulation (TMS) paired with electromyography (EMG) and electroencephalography (EEG).

SECONDARY OUTCOMES:
Change in symptom severity of Suicidal Ideation as measured by by the Scale of Suicide Ideation (SSI) | 2 months
  Scale for Suicide Ideation (SSI); This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas Scale range: 0-38 (total score) Lower scores indicate lower severity of suicidal ideation (i.e., better outcome) Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)
Change in symptom severity of depression as measured by the Hamilton Rating Scale for Depression - 24 | 2 months
  Hamilton Rating Scale for Depression (24-item version); This scale is used to quantify the severity of symptoms of depression Scale range: 0-76 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

OTHER OUTCOMES:
Safety and tolerability as assessed by changes in Blood Pressure (BP) | 1 month
  Assessed through monitoring of systolic and diastolic Blood Pressure (mmHg) on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and tolerability as assessed by changes in Heart Rate (BPM) | 1 month
  Assessed through monitoring of Heart Rate (beats per minute) on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and tolerability as assessed by changes in O2 Saturation | 1 month
  Assessed through monitoring of Oxygen saturation levels on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and Tolerability of IV Ketamine as assessed by monitoring of adverse events | 2 months
  Assessed through monitoring of adverse events, cardiovascular adverse events and/or respiratory distress throughout the trial.
Change in quality of life measures as assessed by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 1 month
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) (12-item version); This scale is used to assess disability over six domains of functioning: cognition, mobility, self-care, getting along with others, participation in society, and life activities.
  Scale range: 12-60 (total score) Lower scores indicate lower disability or loss of function (i.e., better outcome) Higher scores indicate higher disability or loss of function (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Knyahnytska, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Knyahnytska Y, Zomorrodi R, Kaster T, Voineskos D, Trevizol A, Blumberger D. Neural Correlates of the DEEPP (Anti-suicidal Response to Ketamine in Treatment-Resistant Bipolar Depression) Study: Protocol for a Pilot, Open-Label Clinical Trial. JMIR Res Protoc. 2023 Jan 27;12:e41013. doi: 10.2196/41013. PMID 36573651